CLINICAL TRIAL: NCT05774938
Title: QoL After Complex Endovascular Aortic Repair
Status: Recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Rebecka Hultgren, Adjunct professor, Karolinska University Hospital
Other Study IDs: QLEVER
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Quality of Life; Aortic Aneurysm; Aortic Aneurysm, Abdominal
Keywords: Endovascular aneurysm repair; Pararenal aortic aneurysm; Quality of life; Paravisceral aortic aneurysm; Fenestrated endovascular aortic repair; Branched endovascular aortic repair
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard EVAR: Infrarenal abdominal aortic aneurysms treated with standard EVAR off-the-shelf devices.
  Interventions: Procedure: Standard Endovascular aneurysm repair (sEVAR)
- Complex EVAR: Paravisceral aortic aneurysms treated with fenestrated or branched EVAR devices.
  Interventions: Procedure: Complex Endovascular Aneurysm Repair (cEVAR)

INTERVENTIONS:
Procedure: Standard Endovascular aneurysm repair (sEVAR) — Standard EVAR treatment with Medtronic Endurant IIs (Medtronic, Inc. - Minneapolis, Minnesota), Gore Excluder AAA (W. L. Gore & Associates, Inc. - Newark, Delaware), Gore Excluder Conformable AAA (W. L. Gore & Associates, Inc. - Newark, Delaware), Cook Zenith Flex (Cook Medical, Inc. - Bloomington, Indiana).
  Groups: Standard EVAR
Procedure: Complex Endovascular Aneurysm Repair (cEVAR) — Complex EVAR treatment with custom made devices (CMD's) from Cook Medical (Cook Medical, Inc. - Bloomington, Indiana) including fenestrated or branched devices or off-the-shelf T-branch device (Cook Medical, Inc. - Bloomington, Indiana).
  Groups: Complex EVAR

SUMMARY:
The goal of this prospective observational cohort study is to compare health related quality of life in patients with abdominal aortic aneurysms treated by either standard or complex EVAR (endovascular aneurysm repair) devices. The main questions it aims to answer are:

* Compare differences between the physical scores from the preoperative to the postoperative settings between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR)
* To compare long-term physical scores postoperatively between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR) at one year.
* To explore at which time points (if ever) patients treated with standard-EVAR and nonstandard endovascular aortic repair (F-/BEVAR) have restored or normalized physical scores measured by SF-12, measured at 30 days, 6 months, 1 and 3 years.

Participants will be asked to fill out forms pre- and postoperatively with regards to health related quality of life.

The different groups for comparison will be either standard EVAR for infrarenal aortic aneurysms or complex EVAR (fenestrated or branched) for paravisceral aortic aneurysms (PVAAA).

DETAILED DESCRIPTION:
Prospective cohort study with patients planned for elective aortic endovascular repair during a two year time period. The estimated recruitment period is February 2023 - February 2025.

All patients with infrarenal or paravisceral aortic aneurysms planned for treatment with EVAR or F-/BEVAR will be invited to participate in the study at the time of consent of the proposed treatment.

The questionnaires to be filled out will be available online or by paper form. Patient- and aneurysm related variables will be recorded at the time of treatment decision. The endpoint is 3 years of follow up or death. Analysis will be done by both intention-to-treat and per protocol.

The questionnaires to be used are:

* SF-12
* EQ5D
* HADS
* Custom made questionnaire: Education, marital status and need for domestic service

The forms will be filled out at the following intervals:

* Preoperatively (<90 days prior to surgery).
* 30 days postoperatively.
* 6 months postoperatively.
* 12 months postoperatively.
* 36 months postoperatively.

The investigators aim to answer the following research questions:

* Compare differences between the physical scores from the preoperative to the postoperative settings between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR)
* To compare long-term physical scores postoperatively between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR) at one year.
* To explore at which time points (if ever) patients treated with standard-EVAR and nonstandard endovascular aortic repair (F-/BEVAR) have restored or normalized physical scores measured by SF-12, measured at 30 days, 6 months, 1 and 3 years.
* To compare mental scores in SF-12 and HADS postoperatively compared to preoperatively between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR).
* To compare long-term mental scores and HADS-A and HADS-D postoperatively between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR) at one year and three years.
* To evaluate if a decreased function of physical and mental scores in EQ5D or SF-12 should be considered in a preoperative decision model by considering QALYs.
* To compare preoperative physical and mental scores by SF-12 and HADS-A / HADS-D between standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR).
* To compare preoperative and postoperative physical and mental scores by SF-12 and HADS-A / HADS-D between standard EVAR vs de-novo non-standard endovascular aortic repair (F-/BEVAR) vs F-/BEVAR in a previously treated EVAR patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Any age (≥18 years)
* Planned (elective) endovascular treatment by EVAR, FEVAR or BEVAR.
* Patients previously treated by EVAR which are planned for an adjunct fenestrated cuff will not be included in the basic analysis, but included and analysed separately.

Exclusion Criteria:

* Inability to understand and/or respond to the study questionnaires that are in Swedish.
* Inability to provide an informed consent for participation in the study, orally or in writing (This may be due to linguistic or cognitive limitation).
* Participation in other ongoing studies concerning quality of life.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with infrarenal or paravisceral aortic aneurysms planned for treatment with EVAR or F-/BEVAR will be invited to participate in the study at the time of consent of the proposed treatment
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Early physical component score changes after standard or complex EVAR procedure. | 2026
  To compare the difference between the physical scores from the preoperative to the postoperative settings between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR) at 30 days.

SECONDARY OUTCOMES:
Late physical component score changes after standard or complex EVAR procedure. | 2026
  To compare long-term physical scores postoperatively between patients treated with standard EVAR vs non-standard endovascular aortic repair (F-/BEVAR) at one year.
When does physical component scores return to normal after standard or complex EVAR procedures? | 2028
  To explore at which time points (if ever) patients treated with standard-EVAR and nonstandard endovascular aortic repair (F-/BEVAR) have restored or normalized physical scores measured by SF-12, measured at 30 days, 6 months, 1 and 3 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided